CLINICAL TRIAL: NCT01772563
Title: An Open-label Fixed Sequence Trial to Investigate the Potential Drug-drug Interaction of Intravenous Volasertib Co-administered With a P-gp and CYP3A4 Inhibitor (Itraconazole p.o.) in Patients With Various Solid Tumours
Brief Title: Investigation of Potential Drug-drug Interaction of Volasertib With Itraconazole in Patients With Various Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.24; 2011-002367-23 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727; Itraconazole

ARMS (1):
- Volasertib + itraconazole then volasertib (Experimental): Administration of volasertib in combination with itraconazole (Cycle 1) and afterwards alone (Cycle 2 and beyond).
  Interventions: Drug: volasertib; Drug: itraconazole

INTERVENTIONS:
Drug: volasertib — Solution for infusion
Drug: itraconazole — capsules
  Other Names: Orungal®

SUMMARY:
The primary objective of the present study is to investigate the influence of co-administration of itraconazole and volasertib on the pharmacokinetic profile of volasertib without co-administration of itraconazole. Secondary objectives are to investigate safety, tolerability and preliminary therapeutic effects following intravenous administration of volasertib.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed diagnosis of advanced, non resectable and / or metastatic solid tumour, for whom conventional treatment has failed, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment based on the investigator's assessment
2. Male or female
3. Age =>18 and =<70 years
4. Eastern Cooperative Oncology Group (ECOG) performance score =< 2
5. Recovery from Common Terminology Criteria for Adverse Events (CTCAE) Grade >= 2 therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapy (except alopecia)

Exclusion criteria:

1. Serious concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
2. Active infectious disease
3. Viral hepatitis, HIV infection
4. Clinical evidence of active brain metastasis or leptomeningeal disease during the past 6 months
5. Second malignancy currently requiring active therapy (except for hormonal / antihormonal treatment e.g. in prostate or breast cancer)
6. Absolute neutrophil count less than 1,500/mm3
7. Platelet count less than 100,000/mm3
8. Total bilirubin greater than 1.5 mg/dL (> 26 µmol/L, SI unit equivalent)
9. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
10. Serum creatinine greater than 2x upper limit of normal (ULN)
11. QTcF prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).The QTcF will be calculated as the mean of the 3 ECGs taken at screening
12. Female patients with childbearing potential and unwilling to use a medically acceptable method of contraception during the trial and for at least six months after end of active therapy. Woman of childbearing potential (premenopausal female) is defined as the female who is not surgically sterilised by hysterectomy or bilateral tubal ligation or post-menopausal for at least 12 months.
13. Treatment with other investigational drugs or participation in another clinical trial within the past four weeks prior to start of therapy or concomitantly with this trial
14. Chemo-, radio- immuno-, or molecular-targeted cancer-therapy within the past four weeks prior to start of therapy or concomitantly with this trial. This restriction does not apply to steroids, bisphosphonates hormonal / antihormonal treatment (e.g. in prostate or breast cancer).
15. Alcohol abuse more than an average 3 units of alcoholic beverages per day or more than 21 units per week (1 unit equals 0.5 pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) or drug abuse
16. Life expectancy less than 12 weeks
17. Potent CYP 3A4 and P-glycoprotein inhibitors other than the study drug or inducers between one week prior to first drug administration or expected treatment with a respective drug until the last PK sample is collected

    1. Strong CYP 3A4 inhibitors: atazanavir, clarithromycin, indinavir, itraconazole (other then study drug), ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin
    2. CYP 3A4 inducers: carbamazepine, rifampicin
    3. P-gp inhibitors: cyclosporine, erythromycin, itraconazole (other then study drug), ketoconazole, quinidine, phenobarbital salt with quinidine, ritonavir, valspodar, verapamil
    4. P-gp inducers: hypericum perforatum, rifampicin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Hungary (2):
  - PRA Hungary Ltd., Phase I. Clinical Pharmacology Unit, Budapest
  - National Institute of Oncology, Budapest

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lang I, Liu D, Fritsch H, Taube T, Chizhikov E, Liptai B. Potential Drug-Drug Interactions with Combination Volasertib + Itraconazole: A Phase I, Fixed-sequence Study in Patients with Solid Tumors. Clin Ther. 2020 Nov;42(11):2214-2224. doi: 10.1016/j.clinthera.2020.09.015. Epub 2020 Nov 1. PMID 33139055
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was an uncontrolled, open-label, sequential Drug-drug interaction (DDI) trial of volasertib and itraconazole in patients with advanced, non-resectable and/or metastatic solid tumours, for whom conventional treatment had failed or if they were not amenable to established treatment options.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Volasertib + Itraconazole Then Volasertib: Patients were administered from Day-3 to Day 15 of Cycle 1 (cycle duration=21 days) once daily two capsules of 100 milligram (mg) of itraconazole (Orungal®) (total daily dose=200 mg) orally. On Day 1 of Cycle 1 patients were also administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
  On Day 1 of Cycle 2 (cycle duration=21 days) patients were administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
  After Cycle 2 (i.e cycles ≥3): Patients with clinical benefits were administered intravenously on Day 1 of each cycle (cycles ≥3) solution for infusion of volasertib.
Period: Cycle 1
Arm/Group | Volasertib + Itraconazole Then Volasertib
Started | 28
Treated With 300 mg Volasertib | 3
Treated With 250 mg of Volasertib | 25
Completed (Patients continuing to >=Cycle 2) | 24
Not Completed | 4
Not completed — Dose limiting toxicity | 2
Not completed — Progressive disease | 2
Period: Cycle 2 and Beyond
Arm/Group | Volasertib + Itraconazole Then Volasertib
Started (Patients started mono-therapy (Cycle 2 and beyond)) | 24
Treated With 300 mg Volasertib in Cycle 2 | 1
Treated With 250 mg Volasertib in Cycle 2 | 21
Treated With 200 mg Volasertib in Cycle 2 | 1
Completed | 1
Not Completed | 23
Not completed — Progressive disease | 17
Not completed — Refused continuing medication | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients who received at least 1 dose of volasertib. This was the full analysis set; it was mainly used for safety analyses.
Arm/Group | Volasertib + Itraconazole Then Volasertib
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to the Last Quantifiable Drug Plasma Concentration After Dose Administration (AUC0-tz) of Volasertib and Its Metabolite CD 10899
Description: Area under the plasma concentration-time curve over the time interval from zero to the last quantifiable drug plasma concentration after dose administration (AUC0-tz) of volasertib and its metabolite CD 10899 is reported.
Time Frame: 30 minutes before volasertib administration and 1 hour (h), 1.75h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 168h, 336h, 504 h after volasertib administration on Day 1 of Cycle 1 (Volasertib+ Itraconazole) and of Cycle 2 (Volasertib).
Population: Primary pharmacokinetic set (pPKS) 250 mg: All patients in the treated set (TS) who were treated with volasertib 250 mg in Cycle 1 and Cycle 2 and who provided complete pharmacokinetic (PK) measures without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Volasertib+ Itraconazole (Cycle 1): Patients were administered from Day-3 to Day 15 of Cycle 1 (cycle duration=21 days) once daily two capsules of 100 milligram (mg) of itraconazole (Orungal®) (total daily dose=200 mg) orally. On Day 1 of Cycle 1 patients were also administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
- Volasertib (Cycle 2): On Day 1 of Cycle 2 (cycle duration=21 days) patients were administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
Arm/Group | Volasertib+ Itraconazole (Cycle 1) | Volasertib (Cycle 2)
Number analyzed (Participants) | 21 | 21
nanogram*hour/milliliter (ng*h/mL)
  volasertib | 6690 (36.0) | 7140 (55.6)
  CD 10899 | 855 (63.8) | 1130 (58.0)
Statistical Analysis 1: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of Volasertib: AUC0-tz was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 93.63, 90% CI 2-sided [82.07 to 106.81] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV%)=25.1
Statistical Analysis 2: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of CD 10899: AUC0-tz was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 75.77, 90% CI 2-sided [67.830 to 84.632] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV %)=21.0

2. Primary Outcome: Maximum Measured Concentration of Volasertib and Its Metabolite CD 10899 in Plasma (Cmax)
Description: Maximum measured concentration of the analyte (volasertib and its metabolite CD 10899) in plasma (Cmax) is reported.
Time Frame: 30 minutes before volasertib administration and 1 hour (h), 1.75h, 4h, 6h, 8h, 12h, 24, 36h, 48h, 72h, 168h, 336h, 504 h after volasertib administration on Day 1 of Cycle 1 (Volasertib+ Itraconazole) and of Cycle 2 (Volasertib).
Population: Primary pharmacokinetic set (pPKS) 250 mg: All patients in the treated set (TS) who were treated with volasertib 250 mg in Cycle 1 and Cycle 2 and who provided complete pharmacokinetic set (PK) measures without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Volasertib+ Itraconazole (Cycle 1) | Volasertib (Cycle 2)
Number analyzed (Participants) | 21 | 21
nanogram/milliliter (ng/mL)
  volasertib | 328 (46.0) | 414 (53.1)
  CD 10899 | 4.51 (78.4) | 7.10 (63.4)
Statistical Analysis 1: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of volasertib: Cmax was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 79.40, 90% CI 2-sided [64.896 to 97.137] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV %)=39.3
Statistical Analysis 2: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of CD 10899: Cmax was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 63.48, 90% CI 2-sided [55.372 to 72.775] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV%)=26.1

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From 0 to Infinity (AUC0-∞) of Volasertib and Its Metabolite CD 10899
Description: Area under the plasma concentration-time curve over the time interval from 0 to infinity (AUC0-∞) of volasertib and its metabolite CD 10899 is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Volasertib+ Itraconazole (Cycle 1) | Volasertib (Cycle 2)
Number analyzed (Participants) | 21 | 21
nanogram*hour/milliliter (ng*h/mL)
  volasertib | 7360 (38.4) | 7610 (55.5)
  CD 10899 | 1020 (67.1) | 1310 (61.9)
Statistical Analysis 1: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of volasertib: AUC0-∞ was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 97.85, 90% CI 2-sided [87.09 to 109.94] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV %)=22.7
Statistical Analysis 2: Comparison: Volasertib+ Itraconazole (Cycle 1) vs Volasertib (Cycle 2); Statistical analysis of CD 10899: AUC0-∞ was log-transformed prior to fitting an analysis of variance (ANOVA) model. This model included effects for 'treatment' and 'subject'. 90% confidence intervals (CIs) were computed, then back-transformed to the original scale to give the point estimator and interval estimates for the geometric mean ratio (GMR); Test type: Other; Geometric mean ratio (GMR) [%] = 77.42, 90% CI 2-sided [69.001 to 86.871] — GMR (test/reference) i.e. (Volasertib+Itraconazole/ Volasertib). Intra- individual coefficient of variation (gCV %)=22.5

ADVERSE EVENTS:
Time Frame: Volasertib + Itraconazole (Cycle 1) arm: From start of itraconazole administration until 21 days after the administration of volasertib, up to 24 days. Monotherapy Volasertib (Cycle>=2): From start of monotherapy with volasertib (Day 1 of Cycle 2) until 21 days after the last administration of volasertib, up to 2712 days.
Description: Treated set (TS): All patients who received at least 1 dose of volasertib. This was the full analysis set; it was mainly used for safety analyses.
Groups:
- Volasertib + Itraconazole (Cycle 1): Patients were administered from Day-3 to Day 15 of Cycle 1 (cycle duration=21 days) once daily two capsules of 100 milligram (mg) of itraconazole (Orungal®) (total daily dose=200 mg) orally. On Day 1 of Cycle 1 patients were also administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
- Monotherapy Volasertib (Cycle>=2): This group included all patients who were administered volasertib from Cycle 2 onwards.
  On Day 1 of Cycle 2 (cycle duration=21 days) patients were administered intravenously a single dose of 300 mg of solution for infusion of volasertib as a 2 hour (h) infusion. In case of unexpected toxicity the dose of volasertib was to be reduced to 250 mg or 200 mg.
  After Cycle 2 (i.e cycles ≥3): Patients with clinical benefits were administered intravenously on Day 1 of each cycle (cycles ≥3) solution for infusion of volasertib.
Arm/Group | Volasertib + Itraconazole (Cycle 1) | Monotherapy Volasertib (Cycle>=2)
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/24
Serious Adverse Events (participants affected / at risk) | 12/28 | 11/24
Other Adverse Events (participants affected / at risk) | 21/28 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib + Itraconazole (Cycle 1) (N=28) | Monotherapy Volasertib (Cycle>=2) (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 6
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib + Itraconazole (Cycle 1) (N=28) | Monotherapy Volasertib (Cycle>=2) (N=24)
Anaemia (Blood and lymphatic system disorders) | 9 | 9
Leukopenia (Blood and lymphatic system disorders) | 7 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 5
Platelet count increased (Investigations) | 0 | 4
Headache (Nervous system disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT01772563/Prot_000.pdf
  • Statistical Analysis Plan (2014-07-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT01772563/SAP_001.pdf